CLINICAL TRIAL: NCT02274246
Title: GIMIAS® Tool Validation for the Detection of Left Atrium Fibrosis Through Late Enhancement Magnetic Resonance Image Processing. Pattern Determination in a Cohort of Healthy Volunteers
Brief Title: Validation of the Efficacy of the Tool GIMIAS® for the Assessment of Left Atrial Fibrosis in a Group of Healthy Volunteers (RESTORE-HV)
Acronym: RESTORE-HV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RESTORE-HV
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Left Atrial Fibrosis
Keywords: Segmentation; GIMIAS® program; Atrial fibrillation; Left atrial fibrosis; Healthy volunteers
MeSH Terms: conditions — Atrial Fibrillation | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadobutrol (Experimental): Gadobutrol in Healthy volunteers
  Interventions: Drug: gadobutrol

INTERVENTIONS:
Drug: gadobutrol — Gadobutrol administration in healthy volunteers

SUMMARY:
The purpose of this study is to validate the technique for the detection of left atrial fibrosis through segmentation of endocardial and epicardium landmarks of the images obtained with 3 Tgadobutrol-enhanced magnetic resonance with the software GIMIAS® in a cohort of healthy volunteers, without atrial fibrillation or known cardiovascular risk factors.

DETAILED DESCRIPTION:
3D reconstructions obtained by GIMIAS® will be evaluated. Processing images will be carried out by two independent operators, and will calculate the kappa interobserver agreement .

Subsequently, the processed images are compared with images previously obtained in 10 patients with persistent atrial fibrillation adjusted for sex and age. A qualitative visual comparison will be made.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers capable of being subjected to the prespecified tests of the study.
* Healthy volunteers that sign the informed consent after being informed.

Exclusion Criteria:

* Healthy volunteers with:
* A medical history of atrial fibrillation, hypertension or diabetes mellitus.
* A medical history of heart disease, structural, ischemic or arrhythmic.
* A medical history of chronic obstructive pulmonary disease/obstructive sleep apnoea/hypopnoea syndrome
* Sport habits: intense sport activities during three or more hours in a week
* Any assumption that contraindicates the magnetic resonance and/or the use of gadolinium or other contrast mediums, including a medical history of previous allergic or not allergic reactions with the use of gadolinium or other contrast mediums, bronchial asthma or allergic diseases.
* Pregnancy or breast feeding.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with contrast enhancement in left atrium, measured through the reconstruction and processing of late enhancement magnetic resonance images with GIMIAS. | Baseline

SECONDARY OUTCOMES:
Adverse events | 1 week after intervention
Interobserver variability in the generation of segmented images of left atrium, measured through the kappa index. | 1 week after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Barcelona, Spain